CLINICAL TRIAL: NCT02117583
Title: An Open-Label, Randomized, 2-Cohort, Single-Dose, Crossover Study To Estimate The Effects Of Food On Oxycodone Pharmacokinetics Following Oral Administration Of 40 Mg Doses Of Pf 00345439 Formulation K Taken Whole Or After Chewing In Healthy Volunteers
Brief Title: Effects of Food on Oxycodone Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4501039
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: pharmacokinetics; relative bioavailability; food effects; oxycodone
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment B (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment C (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment D (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, taken whole, single dose, under fasting conditions
  Arms: Treatment A
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, taken whole, single dose, under fed conditions
  Arms: Treatment B
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, Chewed, single dose, under fasting conditions
  Arms: Treatment C
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, Chewed, single dose, under fed conditions
  Arms: Treatment D

SUMMARY:
To estimate the effect of food on the pharmacokinetics and relative bioavailability of oxycodone following oral administration of single 40 mg doses of PF 00345439 Formulation K taken whole or after chewing in healthy volunteers. We have described below the two cohorts each with two arms in this crossover study by listing them as four Arms/Groups in order to capture the differences between the cohorts prior to the crossover and after the crossover. 14 participants are planned for the first cohort and 18 participants are planned for the second cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between 18 and 55 years of age

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* Positive urine drug test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Concentration at time 24 hours (C24) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
Plasma Decay Half-Life (t1/2) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4501039&StudyName=Effects%20of%20Food%20on%20Oxycodone%20Pharmacokinetics%20in%20Healthy%20Volunteers